CLINICAL TRIAL: NCT04936256
Title: Evaluation of Binocular Visual Acuity and Refractive Stability in the Alcon Clareon Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Gainesville Eye Associates (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: CB-20-001
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cataract
Keywords: Monofocal IOL; Clareon
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Bilateral implantation of the Clareon monofocal IOL: Clareon monofocal intraocular lens (IOL)
  Interventions: Device: Clareon

INTERVENTIONS:
Device: Clareon — Clareon monofocal intraocular lens (IOL)

SUMMARY:
The objective is to evaluate refractive stability (spherical equivalent change ≤ 0.50D from 1-month to 3-months).

DETAILED DESCRIPTION:
This study is a single-arm, evaluator masked clinical evaluation study of refractive stability, after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 month and 3 months post-operatively. Clinical evaluations will include measurement of bilateral visual acuity, manifest refraction, and defocus curve.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Presenting for uncomplicated bilateral cataract surgery and have an interest in an IOL option
* Gender: Males and Females.
* Age: 50 or older
* Willing and able to provide written informed consent for participation in the study
* Willing and able to comply with scheduled visits and other study procedures.
* Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract)
* Potential postoperative visual acuity of (20/25 Snellen) or better in both eyes

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Irregular astigmatism (e.g. keratoconus)
* Corneal pathology (e.g. scar, dystrophy, pterygium, severe dry eye)
* Previous radial keratotomy, corneal refractive surgery or other corneal surgery (e.g. corneal transplant, DSAEK, lamellar keratoplasty)
* Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
* Diabetic retinopathy
* Macular pathology (e.g. ARMD, ERM)
* History of retinal detachment
* Any patient based on Barrett toric calculator that will have ≥ 0.75D residual astigmatism if Clareon® non-toric IOL is implanted
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity
* Participation in any investigational drug or device trial within the previous 30 days prior to the start date of this trial (or currently participating)

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects ≥50 years of age presenting for cataract surgery who are appropriate candidates for intraocular lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Blehm, MD, Principal Investigator — Gainesville Eye Associates
Locations (1):
- Gainesville Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Started | 31
Completed | 29
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Only subjects who completed the study are included in the baseline analysis.
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Refractive Stability
Description: Refractive stability (spherical equivalent change ≤ 0.50D from 1-month to 3-months)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Diopters (D)
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Number analyzed (Participants) | 29
Diopters (D) | 0.03 [0.028 to 0.041]

2. Secondary Outcome: Binocular Uncorrected Distance Visual Acuity
Description: Binocular uncorrected distance visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Number analyzed (Participants) | 29
logMAR | -0.01 (0.1)

3. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity
Description: Binocular uncorrected intermediate visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Number analyzed (Participants) | 29
logMAR | 0.16 (0.13)

4. Secondary Outcome: Binocular Corrected Distance Visual Acuity
Description: Binocular corrected distance visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Number analyzed (Participants) | 29
logMAR | -0.04 (0.06)

5. Secondary Outcome: Binocular Distance-corrected Intermediate Visual Acuity
Description: Binocular distance-corrected intermediate visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Number analyzed (Participants) | 29
logMAR | 0.16 (0.13)

6. Secondary Outcome: Binocular Defocus Curve
Description: A binocular defocus curve is obtained by measuring visual acuity (logMAR) at different spherical powers (D).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
Number analyzed (Participants) | 29
logMAR
  -4.0 D | 0.90 (0.13)
  -3.5 D | 0.84 (0.14)
  -3.0 D | 0.73 (0.16)
  -2.5 D | 0.64 (0.16)
  -2.0 D | 0.49 (0.16)
  -1.5 D | 0.34 (0.12)
  -1.0 D | 0.20 (0.12)
  -0.5 D | 0.06 (0.11)
  0.0 D | -0.01 (0.11)
  0.5 D | 0.08 (0.09)
  1.0 D | 0.25 (0.12)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Bilateral Implantation of the Clareon Monofocal IOL
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT04936256/Prot_SAP_000.pdf